CLINICAL TRIAL: NCT05442359
Title: The Effect of Nano-Bio Fusion Gingival Gel Versus Natural Healing on the Palatal Wound Healing After Harvesting Free Gingival Graft.
Brief Title: Effect of Nano-Bio Fusion Gel on Palatal Wound Healing After Free Gingival Graft Harvest.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Mahmoud Abdelrehim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8422
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Free Gingival Graft
Keywords: Nano-Biofusion gel; Stent; Palatal Wound
MeSH Terms: interventions — Stents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nano-biofusion gel gingival gel (NBF) (Experimental): Coverage of the free gingival graft area in the palate with stent
  Interventions: Drug: Nano-bio fusion gingival gel
- stent (Active Comparator): Coverage of the free gingival graft area in the palate
  Interventions: Device: stent

INTERVENTIONS:
Drug: Nano-bio fusion gingival gel — Thin coat applied to cover the palate after free gingival graft harvest. A stent will be placed to retain its effect. Patients will receive the gel to be used at home twice daily till 3rd week and once in the 4th week
  Other Names: NBF gingival gel
  Arms: Nano-biofusion gel gingival gel (NBF)
Device: stent — Applied as a palatal stent for palatal wound
  Arms: stent

SUMMARY:
The main aim of soft tissue grafts is to treat mucogingival defects such as exposed root surfaces or augment gingival tissue dimensions. In single or multiple root coverage procedures, autogenous grafts are considered to be the gold standard. where the palate is considered to be the most frequent site for graft harvesting, this procedure is accompanied with complications such as postoperative pain and bleeding. Despite all materials used in the literature, no proven golden standard exits. This study will compare the effect of Nano-Bio Fusion gingival gel versus natural healing with stent as a palatal dressing in the management of wound healing and pain.

DETAILED DESCRIPTION:
In the literature, there are many modalities proposed in an attempt to decrease such complications such as the use of PRF, non-eugenol dressing Coe-pack, medicinal plant extract, hyaluronic acid. Despite all, no proven gold standard exits.

Nano- Bio Fusion gel is a highly functional paste containing (nano vitamin C, nano vitamin E and propolis extract) that was used before as an adjunct to scaling and root planning in the management of chronic periodontitis.

Owing to its natural composition, Vitamin C enhances the synthesis, maturation, secretion and degradation of collagen. Also, propolis extract is mainly composed of flavonoids possessing antimicrobial, anti-inflammatory and now recognized as owning regenerative capacities.

Whereas vitamin E acts as an antioxidant, free radical scavenger, facilitate angiogenesis and epithelialization. Thus, Nano Bio Fusion gel could be tested as a palatal wound dressing aiming to enhance postoperative wound healing and wound re-epithelization.

Palatal Stent will be used in the control group which was previously used in several studies. The choice of the stent was to confirm that any observed effect will be due to the gel only as stent will be used in both groups. Follow up will be over month.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy/controlled patients scheduled for various periodontal or peri-implant plastic surgeries, requiring palatal free gingival graft harvesting, either epithelialized or de-epithelialized.
* Compliant Patients
* Good Oral Hygiene

Exclusion Criteria:

* Uncontrolled systemic diseases
* Pregnancy or lactating females
* Patients with severe gagging reflex
* Patients unwilling to sign an informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | Change in healing from baseline up to 4 weeks
  Assessment of healing using the healing index scale by Landry with scale starting from (1 for very poor healing and 5 excellent healing)

SECONDARY OUTCOMES:
Post-operative Pain Assessment | 14 days
  Visual Analogue Scale (VAS) will be used to evaluate pain with score staring from 0 (minimal pain) to 10(maximum pain)
Post-operative Pain Assessment | 7 days
  Number of analgesics consumption will be recorded by the patient
Patient Satisfaction | Day 30
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Abdelrehim, Bachelor, Principal Investigator — Cairo University, faculty of dentistry; Weam El-Battawy, PHD, Study Director — Cairo University, faculty of dentistry
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelrehim SMM, Elbattawy WA, Ashour OAM. The effect of nano-bio fusion gingival gel versus palatal stent on the palatal wound healing after harvesting free gingival graft: a randomized controlled clinical trial. BDJ Open. 2025 Aug 11;11(1):73. doi: 10.1038/s41405-025-00360-6. PMID 40790022